CLINICAL TRIAL: NCT06669169
Title: A Randomized, Placebo-Controlled, Double-Blind and Multi-Centre Phase II Clinical Trial：Efficacy and Safety of Jia Shen Tablets in the Treatment of Coronary Heart Disease Complicating Chronic Heart Failure (Syndrome of Yang Qi Deficiency With Blood Stasis)
Brief Title: Efficacy and Safety of Jia Shen Tablets in Chronic Heart Failure
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tasly Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TSL-TCM-JSP-Ⅱ
Record Dates: First submitted 2024-10-31; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo group (Placebo Comparator)
  Interventions: Drug: Jia Shen Tablet Placebo
- Low dose group (Experimental)
  Interventions: Drug: Low dose Jia Shen Tablet
- High dose group (Experimental)
  Interventions: Drug: High dose Jia Shen Tablet

INTERVENTIONS:
Drug: Jia Shen Tablet Placebo — Jia Shen Tablet Placebo contains 4 placebo tablets (0.47 g per placebo tablet),take orally, 2 times a day for 12 weeks
  Arms: Placebo group
Drug: Low dose Jia Shen Tablet — Low dose Jia Shen Tablet contains 2 tablets (0.47 g per tablet) and 2 placebo tablets (0.47 g per placebo tablet),take orally, 2 times a day for 12 weeks
  Arms: Low dose group
Drug: High dose Jia Shen Tablet — High dose Jia Shen Tablet contains 4 tablets (0.47 g per tablet),take orally, 2 times a day for 12 weeks
  Arms: High dose group

SUMMARY:
Evaluate the efficacy and safety of Jia Shen Tablets in patients with Chronic Heart Failure.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-79 years, either sex;
* Meet the diagnostic criteria for CHD and CHF;
* Meet the TCM differentiation criteria of yang qi deficiency and blood stasis in CHF;
* Class Ⅱ to Ⅲ for NYHA functional classification;
* Willing to provide written informed consent.

Exclusion Criteria:

* CHF with acute exacerbation or intravenous drug therapy;
* Received cardiac resynchronization therapy (CRT) or other heart failure devices;
* Within 3 months before randomization, acute coronary syndrome（ACS）, stroke or transient ischemic attack（TIA） occurred or received cardiac revascularization (PCI, CABG);
* Plan to undergo cardiac revascularization (PCI, CABG) or cardiac resynchronization therapy (CRT) during the trial period;
* Severe arrhythmias [such as persistent atrial fibrillation, permanent atrial fibrillation, ventricular tachycardia, second-degree type II or higher sinus or atrioventricular block without pacemaker placement, QT interval (QTc) exceeding 480 ms after heart rate adjustment according to Fridericia's formula, or known history or symptoms of long QT syndrome];
* Severe hypertension (systolic blood pressure ≥180mm Hg or diastolic blood pressure ≥110mm Hg) or hypotension (systolic blood pressure < 90 mmHg);
* Heart failure caused by other cardiovascular diseases such as congenital heart disease, severe stenosis or insufficiency of heart valves, cardiomyopathy (e.g. hypertrophic obstructive cardiomyopathy, restrictive cardiomyopathy, dilated cardiomyopathy, alcoholic cardiomyopathy), moderate pericardial effusion, constrictive pericarditis, and infective endocarditis;
* Combined with liver, kidney, hematopoietic system and other serious primary diseases, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) more than 3 times the upper limit of local laboratory normal value, the estimated glomerular filtration rate (eGFR) < 30 ml/min/1.73m2, Blood potassium > 5.5 mmol/L or hemoglobin (Hb) < 90 g/L; Malignant tumors, severe neuroendocrine system diseases and mental diseases;
* Pregnant or lactating;
* Participating in other interventional clinical studies within 1 month before screening;
* Allergic constitution, or allergic to Chinese medicines of Jia Shen Tablets (such as Periploca sepium, salvia miltiorrhiza, etc.);
* The investigator determines that the patient is unable to complete the study or comply with the requirements of the study.

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2025-01-31 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
6-Minutes-Walking-Distance (6MWD): the change from baseline to Week 12. | Baseline and Week 12.

SECONDARY OUTCOMES:
6-Minutes-Walking-Distance (6MWD): the change from baseline to Week 6. | Baseline and Week 6.
NT-proBNP: the change from baseline to Week 6 and 12. | Baseline, Week 6 and 12.
NT-proBNP: the proportion of patients demonstrating a decrease in NT-proBNP level of at least 30%. | Baseline, Week 6 and 12.
Echocardiogram: Measurements will be made of the left ventricle's end diastolic diameter (LVEDD), end diastolic volume (LVEDV), end systolic volume (LVESV), left ventricular ejection fraction（LVEF）, stroke volume (SV), and cardiac output (CO). | Baseline and Week 12.
NYHA functional classification: Measure the percentage of participants whose NYHA functional classification is improved/worsened/unchanged from baseline to Week 6 and 12. | Baseline, Week 6 and 12.
MLHFQ Score: the change from baseline to Week 6 and 12. | Baseline, Week 6 and 12.
  The MLHFQ consists of 21 elements representing varying degrees of impact of HF on health related quality of life. Each item in this questionnaire is scored from 0 (none) to 5 (very much), and the total item score is from 0 (none) to 105 (very much).
Traditional Chinese Medicine（TCM） Syndrome Score: change from baseline to Week 6 and 12. | Baseline, Week 6 and 12.
  There were 3 primary symptoms and 4 secondary symptoms. The state of the tongue and pulse is used to evaluate and score TCM symptoms. The standard of TCM primary symptoms scored as without 0, light 2, medium 4, heavy 6 points. The standard of TCM secondary symptoms scored as without 0, light 1, medium 2, heavy 3 points. Tongue picture and pulse condition did not count.
Dyspnea, weakness and edema: the rate of disappearance of the symptoms (dyspnea, weakness, and edema) from baseline to Week 6 and 12. | Baseline, Week 6 and 12.
Cardiovascular Adverse Events: Incidence of Cardiovascular AEs（cardiovascular death, hospitalization for worsening heart failure, hospitalization for nonfatal myocardial infarction, hospitalization for nonfatal stroke）. | Week 12.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Tianjin University of traditional Chinese, Tianjin, Tianjin Municipality, China